CLINICAL TRIAL: NCT05034055
Title: A Phase 2 Study of Stereotactic Ablative Radiotherapy(SBRT) Followed by Atezolizumab / Tiragolumab in Treatment-naive Patients With Metastatic Non-small Cell Lung Cancer
Brief Title: Study of Stereotactic Ablative Radiotherapy(SBRT) Followed by Atezolizumab / Tiragolumab in Treatment-naive Patients With Metastatic Non-small Cell Lung Cancer
Acronym: SKYROCKET
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4-2021-0891
Record Dates: First submitted 2021-08-27; First posted 2021-09-05 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-09

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — atezolizumab; Tiragolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- atezolizumab / tiragolumab (Experimental): All patients will receive 1200mg atezolizumab administered by IV infusion on Day 1 of each 21-day cycle after completion of stereotactic body radiotherapy (SBRT) for 21(+5) days. No escalations or reductions in the dose of the investigational product will be allowed.Following the administration of atezolizumab, patients will receive 600mg tiragolumab administered by IV infusion on Day 1 of each 21-day cycle. The tiragolumab dose is fixed and is not dependent on body weight.
  Interventions: Drug: atezolizumab / tiragolumab

INTERVENTIONS:
Drug: atezolizumab / tiragolumab — All patients will receive 1200mg atezolizumab administered by IV infusion on Day 1 of each 21-day cycle after completion of stereotactic body radiotherapy (SBRT) for 21(+5) days. No escalations or reductions in the dose of the investigational product will be allowed.Following the administration of atezolizumab, patients will receive 600mg tiragolumab administered by IV infusion on Day 1 of each 21-day cycle. The tiragolumab dose is fixed and is not dependent on body weight.

SUMMARY:
Radiation can induce immunogenic cell death, local release of inflammatory cytokines, and damage associated molecular patterns (DAMPs) resulting in local effects on endothelial cell expression of adhesion receptors, increased immune cell trafficking, and immune cell activation. Dose, fractionation, and volume of radiation can influence immunologic effects in the tumor microenvironment. Nonclinical studies suggest that despite an initial local depletion of lymphocytes, hypofractionated regimens of radiation may be immune activating. Additionally, recent work suggests that standard fractionation and hypofractionation induce expansion of unique immune populations with standard fractionation favoring a myeloid response and hypofractionation driving a lymphoid response that may be more favorable to adaptive anti-tumor immunity. Compared to high doses of radiation, which induce immunogenic cell death, dose-dependent increases of MHC-I and death receptors, moderate fractional doses of 3-10 Gy may be optimal for activating a type I IFN response in tumor cells via a dose-dependent increase in the cytoplasmic leakage of DNA from micronuclei, which activates the cyclic GMP-AMP synthase/stimulator of interferon genes (cGAS/STING) pathway. Extensive experimental evidence indicates that radiotherapy can work in synergy with immunotherapy to generate T cells that reject not only the irradiated tumor but also the metastases outside of the field of irradiation, which offers a rationale for utilizing radiotherapy to enhance response to immunotherapy where tumors are unlikely to respond to immunotherapy alone.

DETAILED DESCRIPTION:
All patients will receive 1200mg atezolizumab administered by IV infusion on Day 1 of each 21-day cycle after completion of stereotactic body radiotherapy (SBRT) for 21(+5) days. No escalations or reductions in the dose of the investigational product will be allowed.Following the administration of atezolizumab, patients will receive 600mg tiragolumab administered by IV infusion on Day 1 of each 21-day cycle. The tiragolumab dose is fixed and is not dependent on body weight.

ELIGIBILITY:
Inclusion Criteria:

1. Age (at the time of informed consent): 20 years and older
2. Subjects with histologically- or cytologically-confirmed advanced or metastatic non-small cell lung cancer according to 8th edition clinical staging system of the American Joint Committee on Cancer before the start of concurrent chemoradiotherapy
3. ECOG Performance Status Score 0 or 1
4. Patient with no prior systemic treatment for advanced or metastatic NSCLC
5. PD-L1 expression 1%
6. Patients with a life expectancy of at least 3 months
7. Patients with measurable disease
8. Patients whose latest laboratory data meet the below criteria within 7 days before enrollment. If the date of the laboratory tests at the time of enrollment is not within 7 days before the first dose of the investigational product, testing must be repeated within 7 days before the first dose of the investigational product, and these latest laboratory tests must meet the following criteria. Of note, laboratory data will not be valid if the patient has received a granulocyte colony-stimulating factor (G-CSF) or blood transfusion within 14 days before testing.

   * White blood cells ≥2,000/mm3 and neutrophils ≥1,500/mm3
   * Platelets ≥100,000/mm3
   * Hemoglobin ≥9.0 g/dL
   * AST (GOT) and ALT (GPT) ≤3.0-fold the upper limit of normal (ULN) of the study site (or ≤5.0-fold the ULN of the study site in patients with liver metastases)
   * Total bilirubin ≤1.5-fold the ULN of the study site
   * Creatinine ≤1.5-fold the ULN of the study site or creatinine clearance (either the measured or estimated value using the Cockcroft-Gault equation) >45 mL/min
9. Women of childbearing potential (including women with chemical menopause or no menstruation for other medical reasons) #1 must agree to use contraception#2 from the time of informed consent until 5 months or more after the last dose of the investigational product, or until 12 months after SBRT completion, whichever is longer. Also, women must agree not to breastfeed from the time of informed consent until 5 months or more after the last dose of the investigational product, or until 12 months after SBRT completion, whichever is longer.
10. Men must agree to use contraception#2 from the start of study treatment until 7 months or more after the last dose of the investigational product, or until 12 months after SBRT completion, whichever is longer.

    * 1. Women of childbearing potential are defined as all women after the onset of menstruation who are not postmenopausal and have not been surgically sterilized (e.g., hysterectomy, bilateral tubal ligation, bilateral oophorectomy). Postmenopause is defined as amenorrhea for ≥12 consecutive months without specific reasons. Women using oral contraceptives, intrauterine devices, or mechanical contraception such as contraceptive barriers are regarded as having childbearing potential.
    * 2. The subject must consent to use any two of the following methods of contraception: vasectomy or condom for patients who are male or female subject's partner and tubal ligation, contraceptive diaphragm, intrauterine device, spermicide, or oral contraceptive for patients who are female or male subject's partner.

Exclusion Criteria:

1. Patients with known driver oncogenes (EGFR, ALK, ROS1)
2. Multiple lesions that cause RT dose beyond normal organ dose constraints
3. Patients with only lesions such as pleural effusion, peritoneal seeding or leptomeningeal metastases that are not suitable for local RT
4. Patients with multiple primary cancers (with the exception of completely resected basal cell carcinoma, stage I squamous cell carcinoma, carcinoma in situ, intramucosal carcinoma, superficial bladder cancer, thyroid cancer or any other cancer that has not recurred for at least 5 years)
5. Patients with current or past history of severe hypersensitivity to any other antibody products
6. Patients with concurrent autoimmune disease or history of chronic or recurrent autoimmune disease
7. Patients with a current or past history of interstitial lung disease or pulmonary fibrosis diagnosed based on imaging or clinical findings. Patients with radiation pneumonitis may be enrolled if the radiation pneumonitis has been confirmed as stable (beyond acute phase) without any concerns about recurrence.
8. Patients with concurrent diverticulitis or symptomatic gastrointestinal ulcerative disease
9. Patients with any metastasis in the brain or meninx that is symptomatic or requires treatment. Patients may be enrolled if the metastasis is asymptomatic and requires no treatment.
10. Patients with pericardial fluid, pleural effusion, or ascites requiring treatment
11. Patients who have experienced a transient ischemic attack, cerebrovascular accident, thrombosis, or thromboembolism (pulmonary arterial embolism or deep vein thrombosis) within 180 days before enrollment
12. Patients with a history of uncontrollable or significant cardiovascular disease meeting any of the following criteria:

    * Myocardial infarction within 180 days before enrollment
    * Uncontrollable angina pectoris within 180 days before enrollment
    * New York Heart Association (NYHA) Class III or IV congestive heart failure
    * Uncontrollable hypertension despite appropriate treatment (e.g., systolic blood pressure ≥150 mmHg or diastolic blood pressure ≥ 90 mmHg lasting 24 hours or more)
    * Arrhythmia requiring treatment
13. Patients with systemic infections requiring treatment
14. Patients who have received systemic corticosteroids (except for temporary use, e.g., for examination or prophylaxis of allergic reactions) or immunosuppressants within 28 days before enrollment (exception with followings: Patients who received acute, low-dose systemic immunosuppressant medication or a one-time pulse dose of systemic immunosuppressant medication (e.g., 48 hours of corticosteroids for a contrast allergy) are eligible for the study)
15. Patients who have undergone surgery under general anesthesia within 28 days before enrollment
16. Patients who have received radiotherapy within 28 days before enrollment, or radiotherapy to bone metastases within 14 days before enrollment
17. Patients with a positive test result for any of the following: HBs antigen, or HCV antibody (except if HCV-RNA negative)
18. Patients with a negative HBs antigen test but a positive test result for either HBs antibody or HBc antibody with a detectable level of HBV-DNA
19. Women who are pregnant or breastfeeding, or possibly pregnant
20. Patients who have received any other unapproved drug (e.g., investigational use of drugs, unapproved combined formulations, or unapproved dosage forms) within 28 days before enrollment
21. Patients judged to be incapable of providing consent for reasons such as concurrent dementia
22. Other patients judged by the investigator or sub-investigator to be inappropriate as subjects of this study

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2021-12 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | up to 5 years after the end of dosing
  The time from curative surgery (no disease) to recurrence/progression/death and From start of osimertinib to documented radiographic relapse/progression by RECIST 1.1 criteria

SECONDARY OUTCOMES:
Objective response rate (ORR) | Screening, After that, performed every 3 months through study completion, an average of 2 years
  according to RECIST 1.1 criteria
Overall survival (OS) | up to 5 years
  Overall survival will be followed continuously while subjects are on the study drug and every 6 months after discontinuation or progression for up to 5 years following the start of therapy either by direct contact (office visits) or via telephone contact, until death, withdrawal of study consent, or lost to follow-up.
durable clinical benefit rate | an average of 2 years
  Clinical Benefit Rate (CBR) are defined as the percentage of patients with advanced or metastatic cancer who have achieved complete response, partial response and stable disease to a therapeutic intervention in clinical trials of anticancer agents.
Adverse event or adverse experience captured | an average of 2 years
  Safety

CONTACTS AND LOCATIONS:
Overall Officials: Byoung Chul Byoung Chul, Principal Investigator — Severance Hospital, Yonsei University Health System
Locations (1):
- Severance Hospital, Yonsei University Health System, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No